CLINICAL TRIAL: NCT02831231
Title: A Phase I, Double-Blind, Randomized, Multiple-Dose, Pilot Study Comparing Xanomeline Administered Alone to Xanomeline Administered in Combination With Trospium Chloride in Normal Healthy Volunteers
Brief Title: Pilot Study Comparing Effects of Xanomeline Alone to Xanomeline Plus Trospium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAR-001
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xanomeline plus placebo (Active Comparator): Drug: Xanomeline tartrate 75 mg TID, for 225 mg total daily dose Placebo, TID
  Interventions: Drug: xanomeline tartrate
- Xanomeline plus trospium (Experimental): Drug: Xanomeline tartrate 75 mg TID, for 225 mg total daily dose Drug: Trospium chloride 20 mg BID, for a 40 mg total daily dose
  Interventions: Drug: xanomeline tartrate; Drug: Trospium chloride

INTERVENTIONS:
Drug: xanomeline tartrate — xanomeline tartrate, 75 mg capsule, TID
  Other Names: LY246708
Drug: Trospium chloride — trospium chloride, over encapsulated 20 mg tablet, BID
  Other Names: Sanctura
  Arms: Xanomeline plus trospium

SUMMARY:
This study is intended to determine whether the addition of trospium chloride to xanomeline tartrate will ameliorate the peripheral cholinergic side effects that have been previously experienced with xanomeline tartrate when administered alone.

DETAILED DESCRIPTION:
In this inpatient study, volunteers will received either xanomeline alone, or xanomeline plus trospium for 7 days. Subjects will report cholinergic side effects daily via visual analog scales, for each of nausea, vomiting, diarrhea, sweating and excessive salivation. Clinician administered scales will also be administered daily for assessment of the same cholinergic side effects.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be postmenopausal (at least 2 years prior to dosing) or agree to use an acceptable form of birth control from screening until 14 days after completion of the study. If on birth control pills, have been on a stable dose for≥12 months.
* Good general health
* Ability to give informed consent and understand verbal instructions
* Willingness to spend 10 days in an in-patient facility

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results. (Subjects with any history of resolved cancer that is >5 years passed can be included.)
* Body Mass Index <18 or > 40 kg/m2
* History of or high risk of urinary retention, gastric retention, or narrow-angle glaucoma
* History of alcohol or drug abuse within the last 24 months, or current abuse as determined by urine toxicology screen
* Clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening
* Has participated in another clinical trial within 90 days prior to the first dose of study medication
* Needs to take any prescription medication besides the investigational product or those specifically noted above.

Use of any vitamins, herbs, supplements, or over the counter medications are excluded within one week of enrollment, and during the course of the trial. Specifically, subjects may not take Benadryl® for one week prior and during the course of the study.

* Use of any tobacco products within the past 30 days
* Previous positive test for HIV 1 and/or 2, or Hepatitis A, B, or C, or a positive test obtained at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Mean weekly maximum composite Visual Analogue Scale (VAS) score (nausea, diarrhea, sweating, salivation and vomiting combined) comparing xanomeline + placebo to xanomeline + trospium | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Biernat, PhD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No